CLINICAL TRIAL: NCT04583293
Title: Long-term Outcomes After Acute Kidney Injury in Coronavirus Disease (COVID-19)
Brief Title: Acute KIDnEy Injury in CoviD-19
Acronym: AIDED
Status: Completed | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UHDB/2020/076
Record Dates: First submitted 2020-10-06; First posted 2020-10-12 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COVID AKI: Participants who were admitted to the hospital with COVID-19 and developed AKI during their hospital stay.
  Interventions: Other: No intervention
- COVID non-AKI: Participants who were admitted to the hospital with COVID-19 and did not develop AKI during their hospital stay.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This study does not involve any intervention or new treatment.

SUMMARY:
This is a prospective observational parallel group cohort study that will aim to recruit 220 participants who were admitted to the hospital with COVID-19 between 1st March 2020 and 30th June 2020 (Group A - 110 participants who had COVID-19 with AKI; Group B - 110 participants who had COVID-19 without AKI). Data from groups A and B will be compared with AKI and non-AKI groups from an existing study database (ARID study, n=1125) who were recruited before the outbreak of the COVID-19 pandemic (recruitment 2013-2016) and who have all completed at least three years of follow up. Participants who have recovered from COVID-19 will be matched for analysis to participants from the ARID study for AKI status, baseline estimated glomerular filtration rate (eGFR) stage, age (± 5 years) and presence of diabetes. Potential participants will receive a letter of invitation along with a comprehensive participant information sheet (PIS).

DETAILED DESCRIPTION:
After the participants have read and understand the PIS, and had sufficient time (at least 24 hours) to consider their participation in this study, the investigators will ask them to sign a consent form, which shows their willingness to take part. The investigators will then collect information from their medical records about their hospital admission with COVID-19, including their age, ethnicity, medical conditions, length of hospital stay, tablets or any other treatments they received, as well as details of their stay in the intensive care unit.

For the two groups - COVID AKI and COVID non-AKI, telephone follow-up with a study questionnaire will be performed at recruitment, 6-9 months and 12-15 months after hospital discharge. The study questionnaire will include the following:

1. Details of any medical event and date of medical event since last study follow-up.
2. Details of any hospital re-admission.
3. Details of current medication.

In addition, at the same time points, participants will be asked to attend their general practitioner surgery or other clinic to have simple clinical measurements (height, weight and blood pressure), blood and urine tests.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients greater or equal to 18 years of age.
2. Swab results positive for SARS-CoV-2.
3. Patients admitted to the hospital for ≥24hrs.

Exclusion Criteria:

1. Paediatric patients as defined by age of <18 years of age.
2. Patients >90 years of age.
3. Swab results negative for SARS-CoV-2.
4. Patients on haemodialysis or peritoneal dialysis, pre-existing CKD stage 5 (eGFR <15ml/min/1.73m2), solid organ transplant.
5. Inability/refusal to give informed consent to participate.
6. Death during the same hospital admission that AKI occurred.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who were admitted to the hospital with COVID-19:
  * Group A: people who had COVID-19 with AKI.
  * Group B: people who had COVID-19 without AKI.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Incidence of kidney disease progression at 12 months. | 12 months after hospital discharge.
  Kidney disease progression will be defined as a decline in estimated glomerular filtration rate (eGFR; ml/min/1.73m2) of ≥30%

SECONDARY OUTCOMES:
Incidence of albuminuria at 6-9 months. | 6-9 months after hospital discharge.
  Albuminuria will be defined as a urine albumin to creatinine ratio (UACR) of >30mg/mmol.
Incidence of albuminuria at 12-15 months. | 12-15 months after hospital discharge.
  Albuminuria will be defined as a urine albumin to creatinine ratio (UACR) of >30mg/mmol.
Incidence of combined kidney disease progression and albuminuria at 6-9 months. | 6-9 months after hospital discharge.
  Combined kidney disease progression outcome of ≥30% decline in eGFR (ml/min.1.73m2) and/or albuminuria (UACR>30mg/mmol).
Incidence of combined kidney disease progression and albuminuria at 12-15 months. | 12-15 months after hospital discharge.
  Combined kidney disease progression outcome of ≥30% decline in eGFR (ml/min.1.73m2) and/or albuminuria (UACR>30mg/mmol).
Factors associated with all-cause mortality at 6-9 months. | 6-9 months after hospital discharge.
  Multi-variable Cox proportional hazards models will be used to assess the factors associated with all-cause mortality
Factors associated with all-cause mortality at 12-15 months. | 12-15 months after hospital discharge.
  Multi-variable Cox proportional hazards models will be used to assess the factors associated with all-cause mortality
Incidence of hospital readmissions at 6-9 months | 6-9 months after hospital discharge.
  Number of hospital readmissions
Incidence of hospital readmissions at 12-15 months | 12-15 months after hospital discharge.
  Number of hospital readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Nitin V Kolhe, Doctor, Principal Investigator — University Hospitals of Derby and Burton NHS Foundation Trust
Locations (1):
- University Hospitals of Derby and Burton NHS Foundation Trust, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No